CLINICAL TRIAL: NCT02560961
Title: Is Kinesio Taping Better Than Placebo Taping for Improving Performance During Unilateral Vertical Jump and Hop Tests? Protocol Study for a Randomized, Placebo-controlled, Double-blind, Clinical Trials.
Brief Title: Is Kinesio Taping Better Than Placebo Taping for Improving Performance During Unilateral Vertical Jump and Hop Tests?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Daniela Ap. Biasotto-Gonzalez, Doctor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Universidade Nove de Julho
Record Dates: First submitted 2015-08-06; First posted 2015-09-25 (Estimated); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Struck by Soccer Ball
Keywords: Kinesio Taping; Soccer; Hop Test; Vertical Jump

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Kinesio Taping protocol - Group A (Experimental): Kinesio Taping (Kinesio Tex Gold®; color: black) will be applied by an experienced, duly trained researcher. The technique described by Kase [1] for activation of the triceps surae on the dominant leg will be employed, with the volunteer in the prone position, maintaining the dominant leg off the cot with hip extension, knee extension and ankle dorsiflexion to maintain the triceps surae in a stretched position. The tape will be applied in a Y shape beginning with the origin of the muscle (femur condyles) without tension (Anchor I), passing over the belly of the muscle (therapeutic region) with 15 to 20% tension and ending near the posterior surface of the heel (Anchor II) without tension.
  Interventions: Other: Kinesio Taping (Kinesio Tex Gold®; color: black)
- Placebo Taping - Group B (Placebo Comparator): Standard white bandaging tape will be applied by the same researcher who placed the tape in Group A. The technique described by Kase [1] for activation of the triceps surae on the dominant leg will be employed, with the volunteer in the prone position, maintaining the dominant leg off the cot with hip extension, knee extension and ankle dorsiflexion to maintain the triceps surae in a stretched position. The tape will be applied in a Y shape beginning with the origin of the muscle (femur condyles) and ending near the posterior surface of the heel.
  Interventions: Other: Placebo Taping

INTERVENTIONS:
Other: Kinesio Taping (Kinesio Tex Gold®; color: black) — Kinesio Taping technique described by Kase for activation of the triceps surae on the dominant leg will be employed, with the volunteer in the prone position, maintaining the dominant leg off the cot with hip extension, knee extension and ankle dorsiflexion to maintain the triceps surae in a stretched position. The tape will be applied in a Y shape beginning with the origin of the muscle (femur condyles) without tension (Anchor I), passing over the belly of the muscle (therapeutic region) with 15 to 20% tension and ending near the posterior surface of the heel (Anchor II) without tension.
  Arms: Kinesio Taping protocol - Group A
Other: Placebo Taping — Standard white bandaging tape will be applied by the same researcher who placed the tape in Group A. The application will be performed the same way as a kinesio taping.
  Arms: Placebo Taping - Group B

SUMMARY:
Introduction: Kinesio taping consists of the attachment of a thin elastic tape over specific muscles, the thickness of which is similar to that of the epidermis. This tape can be stretched to 140% of its original length, which demonstrates greater elasticity in comparison to conventional bandages. According to the creator of this method, Kinesio taping leads to better muscle activation or inhibition, reduces pain, swelling and muscle spasms and prevents muscle injury. Objective: The aim of the proposed study is to compare and analyze the immediate effect of Kinesio taping and placebo taping on performance during unilateral vertical jump and two hop tests by young professional soccer players. Methods: A randomized, placebo-controlled, double-blind, clinical trial will be conducted involving 100 athletes. The volunteers will be submitted to an evaluation of the dominant lower limb using the Single Leg Hop Test and Single Leg Triple Hop Test as well as the evaluation of a unilateral vertical jump on a pressure platform. The athletes will then be randomly allocated to two groups. Group A will receive Kinesio taping of the triceps surae muscle as described by Kase (2003, 2013) and Group B will receive a placebo taping of the same muscle. After 30 minutes, the volunteers will be submitted to the same evaluation tests. Analysis: Intra-group and inter-group analyses of the results will be performed. Statistical tests will be conducted considering a 5% significance level.

DETAILED DESCRIPTION:
Evaluation procedures The consolidated standards of reporting trials (CONSORT) will be used for the proposed randomized clinical trial.

Personal data will be collected using a chart designed by the authors. This chart will contain the following information: name, date of birth, dominant limb, weight and height. Weight and height will be determined using a digital scale (Worker®) and stadiometer (Sanny®), respectively. The dominant limb will be recorded based on the volunteer's answer to a question regarding which leg he would use for a penalty kick. The BMI will be calculated based on weight and height. Individuals with a BMI greater than 25 Kg/m2 or less than 20 Kg/m² will be excluded to standardize the sample.

All volunteers will then undergo the following evaluations:

• Unilateral vertical jump:

The unilateral vertical jump will be used to measure performance, as this movement requires triceps surae strength [9]. The vertical jump will be evaluated using a pressure plate (BIOMEC 400 v1.1® EMG Systems do Brasil) connected to computer (Inter Core 2 Dual®) with 2 GHz and 250 Giga bytes. This system quantifies the distribution of vertical ground reaction force in a static or dynamic position with a sampling frequency of 40 Hz using four force sensors (two anterior and two posterior) capable of supporting 150 Kg. Each sensor stores analog data, which are amplified and converted to digital data interpreted using the Biomec 400® software program (EMG Systems do Brasil). This system records the distribution of force among the four points and changes in body sway in the anteroposterior (Y axis) and mediolateral (X axis) directions. The force plate will be positioned on an even surface. Levelness will be determined by two levels attached to the extremities of the force plate. The volunteer will be instructed to stand on the dominant leg with hands on the hips and jump as high as possible, landing on the same leg. Initially, three jumps will be performed to familiarize the volunteer with the procedure, with a one-minute rest interval between jumps. After a two-minute rest interval, three additional jumps will be performed with a one-minute rest interval between jumps, which will be considered for evaluation. Jump time will be determined using the following formula:

in which h = jump height in meters, t = jump time in seconds and g = acceleration of gravity (9.81 m/s2).

* Single Leg Hop Test Test commonly used to measure functional performance and progression during lower limb rehabilitation programs [10,11,12], with the distance achieved during a single, one-foot hop recorded [11]. For such, the athlete will stand only on the dominant leg behind a line marked on the floor and will hop as far as possible without using the contralateral leg and without losing balance. The distance will be measured with a metric tape from the line marked on the floor to the most proximal point of the heel landing on the floor at the end of the hop . The volunteers will be instructed to keep their hands on their hips throughout the test to reduce the influence of the upper limbs on the performance of the hop test. Initially, three hops will be performed to familiarize the volunteer with the procedure, with a one-minute rest interval between hops. After a two-minute rest interval, three additional hops will be performed with a one-minute rest interval between hops, which will be considered for evaluation.
* Single Leg Triple Hop Test The volunteer will also be positioned on the dominant leg behind the line marked on the floor and will perform three consecutive hops as far as possible without using the contralateral leg and without losing balance. The final distance will be measured with a metric tape from the line marked on the floor to the most proximal point of the heel landing on the floor at the end of the third hop. The volunteers will be instructed to keep their hands on their hips throughout the test to reduce the influence of the upper limbs on the performance of the hop test.

On both hop tests, landing must be made in a stable fashion without touching the contralateral leg or upper limbs to the floor for a hop to be considered valid.

ELIGIBILITY:
Inclusion Criteria:

* Practitioners of soccer aged 15 to 20 years with a body mass index (BMI) within the ideal range (20 to 25 Kg/m2)

Exclusion Criteria:

* History of musculoskeletal injury in the lower limbs in the previous six months and history of surgery on the lower limbs or back in the previous six months

Ages: 15 Years to 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
• Unilateral vertical jump: | 10 minutes
  The volunteer will be instructed to stand on the dominant leg with hands on the hips and jump as high as possible, landing on the same leg. Initially, three jumps will be performed to familiarize the volunteer with the procedure, with a one-minute rest interval between jumps. After a two-minute rest interval, three additional jumps will be performed with a one-minute rest interval between jumps, which will be considered for evaluation.

SECONDARY OUTCOMES:
• Single Leg Hop Test | 15 minutes
  For such, the athlete will stand only on the dominant leg behind a line marked on the floor and will hop as far as possible without using the contralateral leg and without losing balance. The distance will be measured with a metric tape from the line marked on the floor to the most proximal point of the heel landing on the floor at the end of the hop [13]. The volunteers will be instructed to keep their hands on their hips throughout the test to reduce the influence of the upper limbs on the performance of the hop test. Initially, three hops will be performed to familiarize the volunteer with the procedure, with a one-minute rest interval between hops. After a two-minute rest interval, three additional hops will be performed with a one-minute rest interval between hops, which will be considered for evaluation.

OTHER OUTCOMES:
• Single Leg Triple Hop Test | 15 minutes
  The volunteer will also be positioned on the dominant leg behind the line marked on the floor and will perform three consecutive hops as far as possible without using the contralateral leg and without losing balance. The final distance will be measured with a metric tape from the line marked on the floor to the most proximal point of the heel landing on the floor at the end of the third hop [13,14]. The volunteers will be instructed to keep their hands on their hips throughout the test to reduce the influence of the upper limbs on the performance of the hop test.
  On both hop tests, landing must be made in a stable fashion without touching the contralateral leg or upper limbs to the floor for a hop to be considered valid.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Ap Biasotto-Gonzalez, Doctor, Principal Investigator — Universidade Node de Julho